CLINICAL TRIAL: NCT00322829
Title: Development and Optimization of a GBS Micro Total Analysis System (µTAS) Prototype for the Direct Detection of Group B Streptococci in Vaginal/Anal Specimens From Intrapartum Maternity Patients
Brief Title: Development and Optimization of a GBS Diagnostic Test
Status: Completed | Type: Observational
Sponsor: Laval University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Michel G. Bergeron, MD FRCPC, Professor, Laval University
Other Study IDs: 05-0107
Record Dates: First submitted 2006-05-04; First posted 2006-05-08 (Estimated); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Streptococcus Group B
Keywords: Group B Streptococcus, Strepotococcus agalactiae, detection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Vaginal/anal swab samples taken from pregnant women admitted for delivery to the Centre Hospitalier Universitaire de Québec (CHUQ).
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this clinical study is to develop an easily performed test to detect Group B Streptococcus (GBS) in pregnant women at the time of delivery, which would allow health care providers to make an accurate and rapid decision regarding the administration of antibiotics. Administering antibiotics during delivery reduces significantly the likelihood of transmission of GBS, a bacterium that can cause severe life-threatening disease in newborns. Three hundred and twenty pregnant females between 18 to 44 years of age, who are admitted for delivery at the time of consent, will be recruited at the Centre Hospitalier Universitaire de Quebec. Participation involves being observed for 30 minutes. The research nurse will obtain 2 vaginal/anal samples using standard techniques. One sample will be used to detect GBS with the approved BD GeneOhm StrepB assay and the other sample will be used for the development of the new point-of-care rapid detection GBS test.

DETAILED DESCRIPTION:
Group B Streptococcus (GBS), also known as Streptococcus agalactiae, is a gram-positive diplococcus originally known for causing bovine mastitis and was not demonstrated to be a human pathogen until 1938. In the 1970s, GBS emerged as the leading cause of neonatal morbidity and mortality. GBS causes severe invasive disease in newborns. Approximately 80% of infections in young infants occur within the first week of life and are thus designated as early-onset disease. Late-onset infections usually occur in infants between 1 week and 3 months of age. Young infants with invasive GBS disease usually have sepsis or pneumonia but may, though less frequently, present with meningitis, osteomyelitis, or septic arthritis. Bloodstream infections, with or without pneumonia, are the main manifestation of neonatal GBS disease and are observed in approximately 90% of cases, while meningitis occurs in around 10%. Most early-onset disease results from ascending spread of GBS into the amniotic fluid, which leads to neonatal colonization and to invasive disease in some infants. Perinatal transmission of the organism can occur through both ruptured and intact membranes. Transmission from mother to child has been reported to be 29 times higher in GBS-colonized mothers than in noncolonized mothers. The new Centers for Disease Control and Prevention guidelines recommend universal prenatal culture-based screening for GBS colonization in all pregnant women. A more sensitive rapid-screening test for GBS that could accurately detect women who carry GBS at the time of delivery would obviate the need for prenatal screening while reducing the risk associated with the use of intrapartum prophylaxis with antibotics in non-colonized women. The main objective of the study is to develop and optimize a micro TAS prototype for rapid GBS detection directly from vaginal/anal specimens using swabs collected from pregnant women admitted for delivery. It is expected that this diagnostic system can replace the current "gold standard" which is microbiological culture in selective media for determining GBS colonization. Specific objectives of this study include: (1) analytical sensitivity of the micro TAS prototype (number of GBS colony forming units detected per vaginal/anal specimen) will be determined by using prospectively collected vaginal/anal specimens positive for GBS as well as negative vaginal/anal specimens that will be spiked with various numbers of GBS cells; (2) specificity of the micro TAS prototype (ability to detect specifically GBS nucleotide sequences without detecting other microbial species or human sequences) will be determined by using GBS-negative vaginal/anal specimens and; (3) sample analysis and performance of the micro TAS prototype will be compared to clinical samples with FDA-approved BD GeneOhm StrepB assay . Study participants will include 320 pregnant females between 18 to 44 years of age, who are admitted to the Centre Hospitalier Universitaire de Québec for delivery. Participation involves being observed for 30 minutes. The research nurse will obtain 2 vaginal/anal samples using standard techniques. One sample will be used to detect GBS with the approved BD GeneOhm StrepB assay and the other sample will be used for the development of the new point-of-care rapid detection GBS test.

ELIGIBILITY:
Inclusion Criteria:

1. Be admitted for delivery
2. Be able to provide written informed consent

Exclusion Criteria:

1. Have vaginal bleeding
2. Presence of placenta previa
3. Have urgent indication to proceed to immediate delivery
4. Have any condition which in the opinion of the investigator would impose a health risk to the subject or interfere with the evaluation of the GBS diagnostic

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women admitted for delivery at the Centre Hospitalier Universitaire de Québec (CHUQ)
Sampling Method: Non-Probability Sample
Enrollment: 269 (Actual)
Dates: Start 2006-05; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michel G Bergeron, MD, Principal Investigator — Laval University; Fran Rubin, PhD, Study Director — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- Centre Hospitalier de l'Université Laval/ CHUQ, Québec, Canada